CLINICAL TRIAL: NCT03334825
Title: An Enhanced Housing Placement Assistance (EHPA) Program for Homeless Persons Living With HIV/AIDS in New York City
Brief Title: Enhanced Housing Placement Assistance
Acronym: EHPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Department of Health and Mental Hygiene (Other Government)
Responsible Party: Principal Investigator, Ellen Wiewel, Director of Research and Evaluation, New York City Department of Health and Mental Hygiene
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-049
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-09

CONDITIONS: HIV/AIDS; Housing Problems
Keywords: HIV; housing; homelessness
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced housing placement assistance (Experimental)
  Interventions: Other: Enhanced housing placement assistance
- Standard housing placement assistance (Active Comparator)
  Interventions: Other: Standard housing placement assistance

INTERVENTIONS:
Other: Enhanced housing placement assistance — assistance in the rapid (fast-track) acquisition of permanent housing; and participation in a 12-month support services program designed to prevent PLWHA from relapsing into homelessness, with services focused on increasing clients' capacity to live independently and maintain housing stability
  Arms: Enhanced housing placement assistance
Other: Standard housing placement assistance — standard connections to services and housing programs offered by HASA, HOPWA, or Ryan White
  Arms: Standard housing placement assistance

SUMMARY:
Randomized controlled trial of housing placement assistance for homeless persons with HIV

DETAILED DESCRIPTION:
Approximately 800 persons living with HIV/AIDS (PLWHA) reside in HIV emergency single-room-occupancy (SRO) hotels in New York City and do not have the ability to secure permanent housing on their own. The study evaluated a pilot program which fast-tracked PLWHA from HIV emergency SRO hotels into permanent housing. The Enhanced Housing Placement Assistance (EHPA) program had three components: 1) active recruitment of emergency SRO hotel residents with high need for housing; 2) assistance in the rapid (fast-track) acquisition of permanent housing; and 3) participation in a 12-month support services program designed to prevent PLWHA from relapsing into homelessness, with services focused on increasing clients' capacity to live independently and maintain housing stability. Participants were randomly assigned to either 1) EHPA or 2) usual care, which included standard connections to services and housing programs offered by the New York City HIV/AIDS Services Administration (HASA), Housing Opportunities for Persons With AIDS (HOPWA), or Ryan White services, and were followed over twelve months using a questionnaire developed with significant input from the target population of PLWHA residing in emergency SRO hotels.

ELIGIBILITY:
Inclusion Criteria:

* Person living with HIV in New York City
* Residing in an New York City HASA single-adult single-room-occupancy (SRO) hotel

Exclusion Criteria:

* Inability to provide informed consent
* Inability to complete survey in English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen W Wiewel, DrPH, Principal Investigator — New York City Department of Health and Mental Hygiene; Vivian L Towe, PhD, Principal Investigator — RAND

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study team recruited participants onsite at 22 HIV emergency single adult shelters across NYC between April 2012 and April 2013
Period: Overall Study
Arm/Group | Enhanced Housing Placement Assistance | Standard Housing Placement Assistance
Started | 119 | 117
Completed | 112 | 113
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Housing Placement Assistance | Standard Housing Placement Assistance | Total
Number analyzed (Participants) | 119 | 117 | 236
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [42 to 54] | 48 [40 to 54] | 48 [41.5 to 54]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 84 | 90 | 174
  Female | 30 | 21 | 51
  Transgender | 5 | 6 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic Black | 72 | 70 | 142
  Hispanic | 41 | 37 | 78
  Non-Hispanic White | 5 | 10 | 15
  Unknown | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 119 | 117 | 236
Placement in Permanent Housing [Count of Participants; unit: Participants] — Persons were sampled for this study from emergency housing. Therefore, by design, none were placed in permanent housing at baseline.
  Participants | 0 | 0 | 0
Engagement in HIV Care [Count of Participants; unit: Participants] — any reported HIV viral load (VL) or CD4 test within 12 months pre-enrollment Population: One person enrolled in the EHPA arm had baseline interview data but could not be matched with the HIV surveillance registry, which provided laboratory test results indicative of HIV care and viral suppression, so care and suppression characteristics could not be obtained for this one person
  Participants
    number analyzed (Participants) | 118 | 117 | 235
    (all) | 116 | 117 | 233
HIV Viral Suppression [Count of Participants; unit: Participants] — Last viral load is under 200 copies/mL in the 12 months pre-enrollment Population: One person enrolled in the EHPA arm had baseline interview data but could not be matched with the HIV surveillance registry, which provided laboratory test results indicative of HIV care and viral suppression, so care and suppression characteristics could not be obtained for this one person
  Participants
    number analyzed (Participants) | 118 | 117 | 235
    (all) | 33 | 61 | 94

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Placement in Permanent Housing
Description: supportive housing, rental assistance, other non-emergency housing, etc.
Time Frame: 12 months post-enrollment
Population: persons who survived 12 months post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Housing Placement Assistance | Standard Housing Placement Assistance
Number analyzed (Participants) | 112 | 113
Participants | 53 | 37

2. Secondary Outcome: Number of Participants With Engagement in HIV Care
Description: any reported HIV viral load (VL) or CD4 test
Time Frame: 12 months post-enrollment
Population: persons who survived 12 months post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Housing Placement Assistance | Standard Housing Placement Assistance
Number analyzed (Participants) | 112 | 113
Participants | 109 | 110

3. Secondary Outcome: Number of Participants With HIV Viral Suppression
Description: Last viral load is under 200 copies/mL
Time Frame: 12 months post-enrollment
Population: persons who survived 12 months post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Housing Placement Assistance | Standard Housing Placement Assistance
Number analyzed (Participants) | 112 | 113
Participants | 53 | 64

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Enhanced Housing Placement Assistance | Standard Housing Placement Assistance
All-Cause Mortality (participants affected / at risk) | 6/119 | 4/117
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/117
Other Adverse Events (participants affected / at risk) | 0/119 | 0/117

LIMITATIONS AND CAVEATS:
Rates of viral suppression at baseline were unequal between the two study arms, in spite of randomization.

Electronically reported laboratory test data does not distinguish routine vs. acute medical care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs have been employed by the New York City Department of Health and Mental Hygiene. Dr. Towe is no longer at the New York City Department of Health and Mental Hygiene and is currently at RAND Corporation. Any results communications must be cleared by the New York City Department of Health and Mental Hygiene prior to public release.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-04-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03334825/Prot_SAP_000.pdf
  • Informed Consent Form (2012-04-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT03334825/ICF_001.pdf